CLINICAL TRIAL: NCT05636605
Title: Analysis of the Microenvironment of Lung Cancer and Exploration of the Mechanism of Resistance to Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: K2022179
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — tumor tissue, paracancerous tissue, blood, and lymphonodus
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multiomics analysis — Genome, proteomics, single cell RNA sequencing, and space transcriptome sequencing，etc

SUMMARY:
The investigators plan to conduct a multiomics analysis（such as, Genomics, proteomics, single cell RNA sequencing, space transcriptomics）of tumor tissue and blood, aiming at analyzing tumor heterogeneity, mapping the microenvironment map of lung cancer and exploring the mechanism of sensitivity and resistance to anti-PD1/PD-L1 antibodies.

DETAILED DESCRIPTION:
Lung cancer is a highly heterogeneous disease. Cancer cells and cells within the tumor microenvironment together determine disease progression, as well as response to or escape from treatment. Tumor ecosystems are comprised of cancer cells, infiltrating immune cells, stromal cells, and other cell types together with noncellular tissue components, which interact and collectively determine disease progression as well as response to therapy. It is well known that cancer patients elicit very individualized responses to different treatments, demanding better characterization of the whole tumor ecosystem beyond currently applied clinical typing of somatic mutations in cancer cells.

Immune checkpoint blockers (ICBs) have revolutionized the management of patients with lung cancer. Blocking the interaction between the programmed cell death protein 1 (PD-1) receptor and its primary ligand (PD-L1) has demonstrated remarkable anticancer activity, and anti-PD-1/PD-L1 drugs have been approved both as single agents or in combination with cytotoxic chemotherapy. However, most patients receiving anti-PD-1/PD-L1 monoclonal antibodies do not derive benefit. Hence, there is a crucial need to identify reliable predictive biomarkers of the response to anti-PD-1/PD-L1 agents to develop precision medicine for NSCLC immunotherapy as well as to identify novel mechanisms underlying resistance to ICBs.

To map the cell type-specific landscape of cancer cells and their tumor microenvironment in lung cancer, the investigators plan to conduct a multiomics analysis（such as, Genomics, proteomics, single cell RNA sequencing, space transcriptomics）of tumor tissue and blood, aiming at analyzing tumor heterogeneity, mapping the microenvironment map of lung cancer and exploring the mechanism of sensitivity and resistance to anti-PD1/PD-L1 antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology or hemology diagnostics of lung cancer
* Patients have never received any antineoplastic therapy

Exclusion Criteria:

* Within 5 years or at the same time, there are other active malignancies
* Currently participating in interventional clinical research treatment, or received other research drugs or used research devices within 4 weeks before the first administration
* Active autoimmune diseases requiring systemic treatment (such as the use of disease relieving drugs, glucocorticoids or immunosuppressants) occurred within 2 years before the first administration
* The study was receiving systemic glucocorticoid treatment (excluding local glucocorticoids by nasal spray, inhalation or other means) or any other form of immunosuppressive therapy within 7 days before the first administration; Note: It is allowed to use glucocorticoid with physiological dose (prednisone ≤ 10mg/day or equivalent)
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed lung cancer patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate | three years
  Refers to the proportion of patients whose tumor shrinkage reaches a certain amount and remains for a certain period of time, including CR + PR cases
Major Pathologic Response | three-four months
  <10% viable tumor in resected lung and lymph nodes
progression-free survival | three years
  Patients with oncological diseases have a period of time from the start of treatment to the observation of disease progression or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, PhD, Principal Investigator — The Fourth Affiliated Hospital of Zhejiang University
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided